CLINICAL TRIAL: NCT00511927
Title: Observational Study on Prevalence and Prognostic Value of Growth Hormone Deficiency in Patients With Chronic Heart Failure
Brief Title: Growth Hormone Deficiency in Chronic Heart Failure: an Observational Study
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Antonio Cittadini, Associate Professor of Internal Medicine, Federico II University
Other Study IDs: GH Deficiency in CHF
Record Dates: First submitted 2007-08-03; First posted 2007-08-06 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-02

CONDITIONS: Ischemic Heart Disease; Cardiomyopathy; Heart Failure; Growth Hormone Deficiency
Keywords: heart; failure; growth; hormone; igf; dilative; cardiomyopathy
MeSH Terms: conditions — Myocardial Ischemia; Cardiomyopathies; Heart Failure; Dwarfism, Pituitary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sera of the patients at time-points upon recruitment and after 12 months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- GHD: Patients with Growth Hormone Deficiency
- non-GHD: Patients with CHF, without coexisting growth hormone deficiency

SUMMARY:
Aim of this study is to define the possible detrimental effect of a lack of growth hormone, on the well-being and life expectation of patients affected by heart failure.

DETAILED DESCRIPTION:
Growth hormone and its main effector IGF-1 have well-documented roles in the regulation of cardiac and circulatory function. Evidence suggests that GH/IGF-1 exert a beneficial effect on cardiac load, cardiac growth and remodeling, despite their hypertrophying action. Several studies in the last years have demonstrated worse cardiovascular outcomes in adult patients with GH deficiency and/or low levels of IGF-1.

A wide range of alterations in the GH/IGF-1 axis have been described to date in patients with chronic heart failure (CHF): reductions in GH levels, reductions in IGF-1 and a pattern of peripheral resistance to GH, in particular in patients with severe heart failure and cardiac cachexia. Our study hypothesis is that an actual status of GH deficiency coexists with CHF in a large percent of patients, and that it may represent a predictor of worse functional status and possibly of a worse prognosis. Aim of this study is to explore the latter hypothesis, comparing the clinical and functional evolution of patients with CHF and GHD with that of a general CHF population.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Heart Failure: NYHA class II to IV, ACC/AHA stage C/D
* Left ventricular end diastolic diameter >60 mm
* Left ventricular ejection fraction < 40%
* Clinical stability, guideline-oriented top pharmacological therapy
* Informed consent

Exclusion Criteria:

* Active Myocarditis
* Hypertrophic Cardiomyopathy
* Active endocarditis
* Active malignancy
* End stage renal disease
* Severe liver disease (Child B-C)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic heart failure due to left ventricular systolic dysfunction
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2010-07; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
overall survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Cittadini, MD, Study Director — Federico II University; Luigi Saccà, MD, Study Chair — Federico II University
Locations (1):
- III Medicina Interna - Federico II University, Naples, Italy